CLINICAL TRIAL: NCT06125821
Title: Arabic Version Of Henry Ford Hospital Headache Disability Inventory Questionnaire : Cross Cultural Adaptation, Validity, And Reliability
Brief Title: Arabic Version Of Henry Ford Hospital Headache Disability Inventory Questionnaire : Validity, And Reliability
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Ali Mohamed Abd Alghani, principal investigator, Cairo University
Other Study IDs: Arabic Version questionnaire
Record Dates: First submitted 2023-09-28; First posted 2023-11-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire: Arabic Version Of Henry Ford Hospital Headache Disability Inventory Questionnaire : Cross Cultural Adaptation, Validity, And Reliabilit
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
ARABIC VERSION OF HENRY FORD HOSPITAL HEADACHE DISABILITY INVENTORY QUESTIONNAIRE: CROSS-CULTURAL ADAPTATION, VALIDITY, AND RELIABILITY

DETAILED DESCRIPTION:
This questionnaire will be developed to assess the impact of headache on functional and emotional aspects of daily life. The Alpha version of HDI (alpha-HDI) included 40 items, but the newest Beta version (beta-HDI) contains 25 items. The Beta version of HDI, developed by Jacobson (1994) in English, is a generic headache disability questionnaire widely administered in the related research studies.

This questionnaire measures the effect of different medical and rehabilitation treatments on the physical and emotional disabilities in patients with different types of headaches. This generic headache questionnaire is not specific to any headache type. Therefore, HDI will be applied to follow the general consequences of different headache types and to compare different aspects of disability for a variety of headaches. Based on the literature, the original HDI has strong internal consistency/reliability and construct validity. The results of test-retest showed that HDI has an acceptable level of reliability considering the total questionnaire and its subscale scores.

The validity and reliability of the non-English versions of HDI, such as Spanish, have been previously investigated and confirmed. The Arabic researchers and practitioners need valid and reliable tools to measure the emotional and functional states of patients with different headache disorders.

So, This study will be carried out to translate and culturally adapt the HDI questionnaire for administration among the Egyptian patients with headaches. Moreover, This study will assess the validity and reliability of the developed Arabic version of this questionnaire. Creation of questionnaires in different languages must pass through many steps. Questionnaires must be translated, then culturally adapted to the environment in which they will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic primary headache to enter the study.
2. Patients having chronic daily headaches at least 15 days a month.

Exclusion Criteria:

1. Patients with secondary headaches who has underlying serious problems (infection, trauma, tumors, and brain bleedings)
2. Severe psychotic and mental dysfunctions

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In order to select the participants, researchers will examine the patients who referred to the hospital over a 3-month period and selected those diagnosed with chronic primary headache to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Arabic Version Of Henry Ford Hospital Headache Disability Inventory Questionnaire : Cross Cultural Adaptation, Validity, And Reliability | 4 month
  This study will be carried out to translate and culturally adapt the Henry ford inventory questionnaire for administration among the Egyptian patients with headaches.
Arabic Version Of Henry Ford Hospital Headache Disability Inventory Questionnaire : Cross Cultural Adaptation, Validity, And Reliability | 4 month
  This study will assess the validity and reliability of the developed Arabic version of this questionnaire.